CLINICAL TRIAL: NCT07261748
Title: MENA Consensus on Poly-L-Lactic Acid (PLLA) Biostimulator Use in Aesthetic Dermatology
Status: Enrolling by invitation | Type: Observational
Sponsor: Venus Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: PLLA-VenusRC
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Aesthetic Procedures; Cosmetic Techniques; Skin Aging; Rejuvenation
Keywords: Poly-L-lactic acid; PLLA; Biostimulator; Aesthetic dermatology; Collagen biostimulation; MENA region; Delphi study; Expert consensus; Cosmetic injectables; Facial rejuvenation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Expert Panel: A cohort of dermatology and aesthetic medicine experts from the MENA region participating in a Modified Delphi process to develop consensus recommendations on PLLA biostimulator use.

SUMMARY:
This study aims to develop expert consensus on the safe and effective use of poly-L-lactic acid (PLLA) biostimulators in aesthetic dermatology across the Middle East and North Africa (MENA) region. PLLA is a commonly used injectable treatment that stimulates collagen production, but most guidelines come from Western populations and do not address the unique characteristics of Fitzpatrick III-VI skin types, which are predominant in the MENA region.

The study uses a Modified Delphi method, a well-established approach for collecting and refining expert agreement. Dermatologists and aesthetic physicians from MENA countries will participate in two to three online rounds of surveys. In Round 1, experts will answer open-ended questions about indications, contraindications, dilution techniques, safety concerns, anatomical considerations, and training needs related to PLLA. Their responses will be analyzed and converted into structured statements.

In Round 2, experts will rate each statement using a 1-to-9 Likert scale, indicating their level of agreement. Items with high agreement will form part of the final consensus. Statements with uncertain or conflicting ratings may undergo a third round for clarification.

No patients are involved in the study, and no treatments or interventions will be administered. The study collects professional opinions only, and all responses are anonymized during analysis. The final output will be a region-specific clinical guideline to support safer and more standardized PLLA use across the MENA region. Results will be published in peer-reviewed journals and shared with the aesthetic medical community.

DETAILED DESCRIPTION:
Study Overview This study is a non-interventional, observational expert consensus project designed to develop region-specific guidelines for the use of poly-L-lactic acid (PLLA) biostimulators in aesthetic dermatology across the Middle East and North Africa (MENA) region. PLLA is widely used for collagen stimulation and facial rejuvenation, but existing evidence and guidelines are derived primarily from Western populations. Given that Fitzpatrick III-VI skin types dominate the MENA region, and that anatomical, cultural, and safety considerations differ, a structured expert consensus is required to optimize clinical practice.

Study Design

This study uses a Modified Delphi methodology, incorporating principles from the RAND/UCLA Appropriateness Method. The Delphi process includes 2-3 survey rounds:

Round 1 (Qualitative Item Generation):

Experts complete an open-ended questionnaire addressing indications, contraindications, dilution protocols, injection techniques, safety concerns (including risk of papules and PIH), anatomical considerations, combination treatments, follow-up practices, regulatory issues, training requirements, and research priorities. Responses undergo thematic analysis to generate structured candidate statements.

Round 2 (Quantitative Consensus Rating):

The consolidated statements are rated using a 9-point Likert scale (1 = inappropriate, 9 = appropriate). Experts rate each item independently based on clinical relevance, safety, and applicability in MENA populations.

Optional Round 3:

Statements without clear consensus are redistributed with anonymized group statistics for re-rating. This step is used only if needed to refine borderline items.

Expert Panel Selection

Experts will be eligible if they meet at least two of the following:

* ≥5 years of aesthetic practice;
* ≥50 PLLA cases performed;
* Recognized trainer, lecturer, or KOL;
* Publications or academic contributions in aesthetic medicine;
* Active practice within Egypt or other MENA countries. Panel size will be 15-25 experts, ensuring geographic, academic, and experiential diversity.

Consensus Definitions

The study follows RAND/UCLA criteria:

* Consensus (Appropriate): Median 7-9 AND Disagreement Index (DI) < 1.0
* Consensus (Inappropriate): Median 1-3 AND DI < 1.0
* No Consensus: Median 4-6 OR DI ≥ 1.0
* Items with near-consensus may undergo a third Delphi round. Data Collection Tools

VRC-developed materials include:

* Full A-L Likert questionnaire
* Fillable PDF form
* Online REDCap/Google Forms instrument
* Round-2 survey booklet
* Excel master sheet for response tracking Statistical Analysis For each item, the following will be calculated: median, interquartile range, interpercentile range (IPR), IPR adjusted for symmetry (IPRAS), and the Disagreement Index. Items will be categorized by agreement level and summarized for publication. Subgroup analyses (e.g., GCC vs North Africa) may be performed.

Ethical Considerations This study does not involve patients, clinical interventions, or personal health information. Participation is voluntary. Expert responses are anonymized. No foreseeable risks are associated with participation, and the study qualifies as minimal-risk, non-interventional research.

Outcomes and Dissemination The primary outcome is a set of consensus-based, region-specific recommendations for PLLA use in aesthetic practice. Secondary outcomes include identification of training standards and research priorities. Results will be disseminated through peer-reviewed publications, conference presentations, and a VRC-branded clinical guideline.

ELIGIBILITY:
Inclusion Criteria:

* Board-certified dermatologist or plastic surgeon OR physician practicing aesthetic medicine.
* Minimum of 5 years of clinical experience OR ≥50 documented PLLA cases.
* Practicing within Egypt or the Middle East and North Africa (MENA) region.
* Willingness to participate in Delphi rounds and provide expert ratings.
* Ability to read and respond to surveys in English.

Exclusion Criteria:

* Inability or unwillingness to complete Delphi rounds.
* Lack of clinical experience with PLLA.
* Industry representatives without direct clinical practice.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A purposively selected group of dermatology and aesthetic medicine experts from Egypt and the broader MENA region. Participants are clinicians with significant experience using poly-L-lactic acid (PLLA) biostimulators and are invited to contribute to a structured Modified Delphi process to develop regional consensus recommendations.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Achievement of Consensus on PLLA Clinical Practice Statements | 6-12 weeks
  The primary outcome is the proportion of Delphi statements reaching consensus among expert panelists. Consensus is defined using RAND/UCLA criteria: a median rating of 7-9 on a 9-point Likert scale with a Disagreement Index (DI) < 1.0. Statements will be categorized as "consensus appropriate," "consensus inappropriate," or "no consensus."

SECONDARY OUTCOMES:
Expert Rating Distribution Across PLLA Practice Domains | 6-12 weeks
  Distribution of Likert scores (1-9) for each PLLA practice statement across domains (patient selection, dilution, technique, safety, anatomy, consent, combinations, ultrasound use, follow-up, regulatory, training, research priorities). Medians, interquartile ranges, and DI will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Venus Research Center, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Delphi studies do not collect patient data, medical records, biological samples, or identifiable clinical information. Experts only give opinions, not "IPD." Their responses are anonymized, and sharing identifiable expert-level responses is not required and often discouraged